CLINICAL TRIAL: NCT06151886
Title: Experiences and Challenges in Life-dependent Home Mechanical Ventilation - a Part of the Air For Life Project
Brief Title: Life-dependent Home Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anne Kathrine Staehr-Rye, Principal investigator, clinical associate professor, Rigshospitalet, Denmark
Other Study IDs: J-23039527
Record Dates: First submitted 2023-09-06; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Ventilator Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients
- Relatives
- Trained respiratory patient caregiver

SUMMARY:
In Denmark, life-dependent home-mechanical ventilation (HMV) is given under the surveillance of a specifically trained respiratory patient caregiver (tPCG). The HMV can be invasive through a tracheostomy or non-invasive via a mask.

The purpose of this study is to uncover experiences and challenges associated with having a trained respiratory patient care giver (tPCG) to surveil home-mechanical ventilation (HMV) from the perspective of the patients and their families and to gather information about the expirence of working in a home as a tPCG

ELIGIBILITY:
Inclusion Criteria:

Patient Age > 18 years Has trained patient care givers to surveil the respiratory treatment and working on the responsibility of the Respiratory Center East

Parent Age > 18 years Has a child less than 18 years old with tPCG, working on the responsibility of the Respiratory Center East, to surveil the home-mechanical ventilation

Other relative:

Age > 18 years Involved in the treatment or support of a relative with tPCG, working on the responsibility of the Respiratory Center East, to surveil the home-mechanical ventilation

Trained patient caregivers (tPCG) Age > 18 years Employed by an external agency or by the patient (BPA) to surveil home-mechanical ventilation Certified as tPCG working on the responsibility of the Respiratory Center East

Exclusion Criteria:

* No informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients assigned with a trained patient care giver to surveil the respiratory treatment (invasive and noninvasive mechanical ventilation) and working on the responsibility of the Respiratory Center East, their relatives as well as trained respiratory patient caregivers working on the responsibility of the Respiratory Center East
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Severe respiratory insufficiency questionnaire | Assessed within the last 7 days
  The patients will be asked to fullfill the questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesia, Pain and REspiratory Support, Glostrup Municipality, Denmark